CLINICAL TRIAL: NCT00889447
Title: Screening Evaluation for Studies of COPD
Brief Title: Screening Evaluation for Studies of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00013323; 1P50HL084945 (NIH)
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research is being done to study mechanisms of progression of COPD and to develop treatments for it. The investigators are doing the present study to identify people age 40 and older with mild to moderate COPD who will qualify for such studies to include in a database. The study will include establishing a screening evaluation or characterization of the following two studies:

* Emphysema Progression in COPD- Losartan's Effects on Airway Parameters - NA_00009980
* Sleep-Related Physiology and Inflammation in Chronic Obstructive Pulmonary Disease - NA_00001771

DETAILED DESCRIPTION:
This is a program to recruit and screen participants for clinical trials or more detailed observational studies of COPD. There are no interventions or comparative results to be published from this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years and older, either sex
* Mild to moderate COPD (FEV1/Forced vital capacity (FVC) ratio ≤ 0.70, FEV1 30-70% predicted, Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥35% predicted)
* On stable maintenance therapy for 2 months
* Current or former smoker (patient report of at least a 10 pack-year history)
* Ability to understand and willingness to sign consent documents

Exclusion Criteria:

* COPD exacerbation requiring treatment within past 6 weeks
* Untreated arterial hypertension (systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg)
* Decompensated heart failure
* Myocardial infarction within past 3 months or ever
* Evidence of interstitial, occupational or chronic infectious lung disease
* Renal dysfunction
* Supplemental oxygen > 2 liters/m at rest
* Failure to keep screening appointments

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both Male and Female 40 years and older
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Establish a screening evaluation or characterization | Determined during screening clinical visit
  We are doing the present study to identify people to include in a database who are age 40 and older with mild to moderate COPD and who will qualify for studies of COPD. The study will include establishing a screening evaluation or characterization for the following three studies.
  * Emphysema Progression in COPD- Losartan's Effects on Airway Parameters - NA_00009980
  * Sleep-Related Physiology and Inflammation in Chronic Obstructive Pulmonary Disease - NA_00001771
  * Genetic Epidemiology of Chronic Obstructive Pulmonary Disease - NA_00011524

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Diette, MD,MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States